CLINICAL TRIAL: NCT04471623
Title: Decentralized Trial in Atrial Fibrillation Patients (DeTAP): Validation of a Combined Digital Health Technology Approach to Fully Decentralize an Intervention to Administer, Promote, and Track Oral Anticoagulant Therapy
Brief Title: Decentralized Trial in Atrial Fibrillation Patients
Acronym: DeTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rajesh Dash, MD PHD, Associate Professor of Cardiovascular Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 57019
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DeTAP Study App and Home Devices (Experimental): Monitoring of OAC administration, OAC adherence, and clinical status through combined decentralized technologies
  Interventions: Behavioral: Use of DeTAP App and Home Devices

INTERVENTIONS:
Behavioral: Use of DeTAP App and Home Devices — DeTAP App (data collection, televisit function, information and reminders), Bluetooth-connected 6-lead home (electrocardiogram) EKG device, Bluetooth-connected blood pressure (BP) cuff

SUMMARY:
The purpose of this study is to validate an approach to decentralize, or virtualize, the clinical trial experience for enrolled subjects, through the coordinated use of multiple digital health and telehealth technologies. The study aims to validate the feasibility, acceptability and best practices of coordinating/integrating several individual digital health technologies to achieve execution of high compliance, cost-efficient, and scientifically sound clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Atrial Fibrillation documented (health record diagnosis or EKG) within the past year and taking an oral anticoagulant (OAC) medication for stroke prevention
* Uses a smart phone daily and is willing to use apps and home devices for the study
* Agreeable to use a Televisit method to conduct all study visits from trial team

Exclusion Criteria:

* Active angina, stable or unstable, requiring urgent cardiovascular functional risk stratification (stress testing or catheterization) or intervention. Or has congestive heart failure that is not compensated or in which the subject is not euvolemic, as determined by the treating MD
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.
* Does not speak English

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Engagement with study protocol | 6 months
  Composite endpoint of:
  * % daily OAC adherence
  * % Completion of telehealth visits
  * % Completion of lab test
  * % Survey completion
Effectiveness of notifications | 6 months
  Composite endpoint of:
  * Time from App-based survey notification to completion
  * Time from App-based lab reminder notification to lab collection
  * Time from App-based home vital sign/EKG reminder notification to vital sign/EKG collection

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Dash, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] K Josan, A Touros, C Petlura, V Parameswaran, U Grewal, M Senior, T Viethen, H Mundl, C Seninger, J Luithle, K Mahaffey, M Turakhia, R Dash, Validation of a pandemic-proof, decentralized cardiovascular trial: scalable design produces rapid recruitment, high engagement and protocol adherence in DeTAP (Decentralized Trial in Afib Patients), European Heart Journal, Volume 42, Issue Supplement_1, October 2021, ehab724.3177, https://doi.org/10.1093/eurheartj/ehab724.3177
- [Result] Sarraju A, Seninger C, Parameswaran V, Petlura C, Bazouzi T, Josan K, Grewal U, Viethen T, Mundl H, Luithle J, Basobas L, Touros A, Senior MJT, De Lombaert K, Mahaffey KW, Turakhia MP, Dash R. Pandemic-proof recruitment and engagement in a fully decentralized trial in atrial fibrillation patients (DeTAP). NPJ Digit Med. 2022 Jun 28;5(1):80. doi: 10.1038/s41746-022-00622-9. PMID 35764796